CLINICAL TRIAL: NCT03159806
Title: Optimising the Recovery of Kidney Function Markers Using a CE-marked Intravenous Microdialysis Probe
Brief Title: Detecting Markers of Kidney Function With Intravenous Microdialysis
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Accunea Ltd. (Industry)
Collaborators: Hammersmith Hospitals NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: MD001
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples retained as per hospital lab protocol, microdialysis samples retained until analysis then discarded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Outpatients: Attendees at the nephrology outpatient clinic at Hammersmith Hospital will be invited to take part in microdialysis sampling
  Interventions: Device: Microdialysis sampling

INTERVENTIONS:
Device: Microdialysis sampling — Insertion of CE-marked intravenous microdialysis catheter, use of CE-marked microdialysis pump to collect intravenous microdialysis samples

SUMMARY:
Patients will be invited to participate from an outpatient nephrology clinic at Hammersmith Hospital. They will have a microdialysis catheter inserted into a peripheral vein and connected to a sampling system. The samples will be sent for analysis in the hospital laboratory. All medical devices to be used are already CE-marked and approved for these purposes.

DETAILED DESCRIPTION:
Patients attending Professor Tam's outpatient clinic will be invited to participate in the study. After time to read the relevant protocol and consent form, and agreeing to proceed, a patient will be taken to a separate room in the outpatient department by Dr. Robert M. Learney.

In this room, the patient will have a suitable vein identified on the forearm or back of the hand. Dr. Learney will then insert a venous cannula into the vein with aseptic technique, secure it in place, and then draw a 3-5mL preliminary blood sample for creatinine and potassium analysis in the hospital lab. Outpatients attending the nephrology department would have one blood test for these biochemicals (and others) taken as part of routine care anyway. This sampling would replace the routine blood test for this attendance.

Dr. Learney will then insert a single-use type 67 intravenous microdialysis catheter into the venous cannula, attach a sampling vial to the outlet of the catheter, and a pump for delivering a sterile saline solution to the inlet of the catheter. All devices and liquids are CE-marked and licensed for human use. Half of the 20 patients in the study will have a short 1cm microdialysis catheter inserted, and half will have a longer 2cm microdialysis catheter inserted.

The pump will be started at a flow rate of 2 microlitres per minute, and 50 microlitres of sample will be collected over the next 25 minutes. The patient will be free to walk around and/or read a book, but must return at the end of 30 minutes for the sample vial to be exchanged for a new one. At this point the pump flow rate will be adjusted down to 1 microlitre per minute by turning a small dial on the side. The patient will be free again for the next 50 minutes to produce the next 50 microlitres of sample. The sample vial will be exchanged again at this point, and the flow rate adjusted down one final time to 0.5 microlitres per minute for 100 minutes to collect a final 50 microlitres of sample.

After this final experiment, the patient will have the microdialysis catheter removed from the cannula for inspection and disposal. A final 3-5mL blood sample will be withdrawn from the cannula, and if this is not possible then it will be taken from a different visible vein. These first and last blood draws ensure that the baseline levels of the two chemicals of interest have not changed significantly during the three hours of the experiment.

All samples collected in this experiment will be assayed in the hospital laboratory for the biochemicals of interest.

ELIGIBILITY:
Inclusion Criteria:

* Attending nephrology outpatient clinic
* Aged 18-85
* Able to spare 3.5 hours to participate in study

Exclusion Criteria:

* Lacks capacity to consent
* Unable to consent in English
* No visible peripheral veins

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal cross-section of adults attending outpatient nephrology clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Recovery of biochemicals of interest | 6 months
  Calculation of optimal microdialysis settings for recovery of specific biochemicals by intravenous microdialysis

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Tam, MBBChir PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stjernstrom H, Karlsson T, Ungerstedt U, Hillered L. Chemical monitoring of intensive care patients using intravenous microdialysis. Intensive Care Med. 1993;19(7):423-8. doi: 10.1007/BF01724886. PMID 8270725